CLINICAL TRIAL: NCT03305146
Title: Study of Feasibility and Diagnostic Profitability of Intra-cyst Fluid Molecular Biology Analysis in Pancreatic Cyst Tumors.
Brief Title: Feasibility of Molecular Biology in Pancreatic Cyst Tumors
Acronym: CYST-GEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Collaborators: Ramsay Générale de Santé (Other)
Responsible Party: Principal Investigator, Arthur Laquiere, Principal Investigator Dr Arthur LAQUIERE, Hospital St. Joseph, Marseille, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01399-42
Record Dates: First submitted 2017-06-14; First posted 2017-10-09 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Cyst; Pancreas Cyst; Serous Cystadenoma; Mucinous Cystadenoma; IPMN
MeSH Terms: conditions — Pancreatic Cyst; Cystadenoma, Serous; Cystadenoma, Mucinous

STUDY DESIGN:
Intervention Model Description: First 20 patients for pilot study to test the feasibility of the molecular analysis then 120 patients to continue the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): For inoperable patients with indeterminate cystic lesions of the pancreas,a EUS FNA will be performed and molecular biology analysis of pancreatic intra-cyst fluid collected by EUS FNA will be performed.
  For operable patients, after the pancreatic surgery, molecular biology analysis of extemporaneous pancreatic tissue specimen biopsy will be conducted.
  Interventions: Genetic: Molecular biology analysis of pancreatic intra-cyst fluid

INTERVENTIONS:
Genetic: Molecular biology analysis of pancreatic intra-cyst fluid — The EUS FNA will be performed according to the Francophone Club of Echo Endoscopy recommendations.
  For molecular biology technique, the samples will be processed within the UMR_S910 unit. Nucleic acids will be extracted from the intra-cystic fluid or, for post-operative patients, from a resected specimen that will be collected into a tube containing a nucleic acid stabilization solution (Allprotect Tissue reagent, Qiagen).
  The nucleic acids will be extracted and then sequenced. The sequencing technology chosen (HaloPlexHS, Agilent) allows a detection close to 1% in allelic frequency. This new technical approach that links high sensitivity and specificity is also suitable with degraded and/or low-volume ( <50ng) DNA.

SUMMARY:
The main objective of the study is to compare the diagnostic accuracy of intra-cystic fluid DNA molecular analysis to standard diagnostics.

The secondary objective of the study is to evaluate the feasibility of intra-cystic fluid DNA molecular analysis.

DETAILED DESCRIPTION:
Multicenter study to determinate the feasibility of intra-cystic fluid DNA molecular analysis in patients with suspected cystic tumours of pancreas in whom EUS FNA is clinically indicated.

Morphological criteria obtained by MRI and computerised tomography (tumor characterization (size, metastases presence, dilatation of bile ducts), etiologic diagnosis, serious symptoms), biological exams (biomarkers), cytological analysis will lead to a diagnosis and a treatment.

The goal of this study is to compare this standard diagnostic modalities to diagnosis obtained by intra-cystic fluid DNA molecular analysis.

Is the DNA molecular analysis improve the diagnosis accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years of age, male or female
* Cystic tumor of the pancreas requiring a puncture under endoscopic control to determine the etiologic diagnosis and gravity.

Exclusion Criteria:

* Doubts regarding the etiological diagnosis of the pancreatic cyst
* Contraindications for the realization of a high digestive endoscopy
* Haemorrhagic disorder, haemostasis and coagulation disorder (TP <60%, TCa> 40 sec and platelets <60000 / mm3).
* AVK, AOD and AAP cannot be stopped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between gene mutations found into the pancreatic cystic tumor fluid to gene mutations found into tissue specimen | 10 days
  The nucleic acids of the samples will be extracted and then sequenced on a panel of about 70 genes implicated in the pancreatic tumorigenesis and targeting RAS, MAPK, AKT, JAK-STAT, WNT, TGFB, TP53 and Repair BRCA, ATM. The selected sequencing technology (HaloPlexHS ®, Agilent) will be used. A comparison of the molecular profiles between the cystic fluid and the surgical specimen will be carried out and then confronted with the pathology, biological, radiological and clinical characterization

SECONDARY OUTCOMES:
Evaluate the feasibility of the molecular biology analysis of the pancreatic cystic tumor fluid to distinguish the pancreatic cysts. | up to 6 months
  The nucleic acids of the samples will be extracted from the different cyst fluids and then sequenced. A comparison of the molecular profiles between the different cystic fluids will be carried out and then confronted with the pathology, biological, radiological and clinical characterization

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Laquière, MD, Principal Investigator — French Society of Digestive Endoscopy
Locations (11):
- France (11):
  - Clinique de Bercy, Charenton-le-Pont
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hopital Mermoz, Lyon
  - Hopital Europeen, Marseille
  - Hopital Saint Joseph, Marseille
  - Chu La Timone, Marseille
  - CHU NANTES Institut des Maladies de l'Appareil Digestif, Nantes
  - Chu L'Archet 2, Nice
  - Hopital Saint Joseph, Paris
  - Centre Hospitalier Jacques Lacarin, Vichy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KS, Sekhar A, Rofsky NM, Pedrosa I. Prevalence of incidental pancreatic cysts in the adult population on MR imaging. Am J Gastroenterol. 2010 Sep;105(9):2079-84. doi: 10.1038/ajg.2010.122. Epub 2010 Mar 30. PMID 20354507
- [Background] Farrell JJ, Fernandez-del Castillo C. Pancreatic cystic neoplasms: management and unanswered questions. Gastroenterology. 2013 Jun;144(6):1303-15. doi: 10.1053/j.gastro.2013.01.073. PMID 23622140
- [Background] Terris B, Ponsot P, Paye F, Hammel P, Sauvanet A, Molas G, Bernades P, Belghiti J, Ruszniewski P, Flejou JF. Intraductal papillary mucinous tumors of the pancreas confined to secondary ducts show less aggressive pathologic features as compared with those involving the main pancreatic duct. Am J Surg Pathol. 2000 Oct;24(10):1372-7. doi: 10.1097/00000478-200010000-00006. PMID 11023098
- [Background] Crippa S, Fernandez-Del Castillo C, Salvia R, Finkelstein D, Bassi C, Dominguez I, Muzikansky A, Thayer SP, Falconi M, Mino-Kenudson M, Capelli P, Lauwers GY, Partelli S, Pederzoli P, Warshaw AL. Mucin-producing neoplasms of the pancreas: an analysis of distinguishing clinical and epidemiologic characteristics. Clin Gastroenterol Hepatol. 2010 Feb;8(2):213-9. doi: 10.1016/j.cgh.2009.10.001. Epub 2009 Oct 14. PMID 19835989
- [Background] Marchegiani G, Mino-Kenudson M, Sahora K, Morales-Oyarvide V, Thayer S, Ferrone C, Warshaw AL, Lillemoe KD, Fernandez-Del Castillo C. IPMN involving the main pancreatic duct: biology, epidemiology, and long-term outcomes following resection. Ann Surg. 2015 May;261(5):976-83. doi: 10.1097/SLA.0000000000000813. PMID 24979607
- [Background] Tanaka M, Fernandez-del Castillo C, Adsay V, Chari S, Falconi M, Jang JY, Kimura W, Levy P, Pitman MB, Schmidt CM, Shimizu M, Wolfgang CL, Yamaguchi K, Yamao K; International Association of Pancreatology. International consensus guidelines 2012 for the management of IPMN and MCN of the pancreas. Pancreatology. 2012 May-Jun;12(3):183-97. doi: 10.1016/j.pan.2012.04.004. Epub 2012 Apr 16. PMID 22687371
- [Background] Brugge WR, Lewandrowski K, Lee-Lewandrowski E, Centeno BA, Szydlo T, Regan S, del Castillo CF, Warshaw AL. Diagnosis of pancreatic cystic neoplasms: a report of the cooperative pancreatic cyst study. Gastroenterology. 2004 May;126(5):1330-6. doi: 10.1053/j.gastro.2004.02.013. PMID 15131794
- [Background] Serikawa M, Sasaki T, Fujimoto Y, Kuwahara K, Chayama K. Management of intraductal papillary-mucinous neoplasm of the pancreas: treatment strategy based on morphologic classification. J Clin Gastroenterol. 2006 Oct;40(9):856-62. doi: 10.1097/01.mcg.0000225609.63975.6f. PMID 17016145
- [Background] Bournet B, Kirzin S, Carrere N, Portier G, Otal P, Selves J, Musso C, Suc B, Moreau J, Fourtanier G, Pradere B, Lazorthes F, Escourrou J, Buscail L. Clinical fate of branch duct and mixed forms of intraductal papillary mucinous neoplasia of the pancreas. J Gastroenterol Hepatol. 2009 Jul;24(7):1211-7. doi: 10.1111/j.1440-1746.2009.05826.x. Epub 2009 May 19. PMID 19476563
- [Background] Sugiyama M, Izumisato Y, Abe N, Masaki T, Mori T, Atomi Y. Predictive factors for malignancy in intraductal papillary-mucinous tumours of the pancreas. Br J Surg. 2003 Oct;90(10):1244-9. doi: 10.1002/bjs.4265. PMID 14515294
- [Background] Kanno A, Satoh K, Hirota M, Hamada S, Umino J, Itoh H, Masamune A, Asakura T, Shimosegawa T. Prediction of invasive carcinoma in branch type intraductal papillary mucinous neoplasms of the pancreas. J Gastroenterol. 2010 Sep;45(9):952-9. doi: 10.1007/s00535-010-0238-0. Epub 2010 Apr 10. PMID 20383536
- [Background] Crippa S, Salvia R, Warshaw AL, Dominguez I, Bassi C, Falconi M, Thayer SP, Zamboni G, Lauwers GY, Mino-Kenudson M, Capelli P, Pederzoli P, Castillo CF. Mucinous cystic neoplasm of the pancreas is not an aggressive entity: lessons from 163 resected patients. Ann Surg. 2008 Apr;247(4):571-9. doi: 10.1097/SLA.0b013e31811f4449. PMID 18362619
- [Background] Cizginer S, Turner BG, Bilge AR, Karaca C, Pitman MB, Brugge WR. Cyst fluid carcinoembryonic antigen is an accurate diagnostic marker of pancreatic mucinous cysts. Pancreas. 2011 Oct;40(7):1024-8. doi: 10.1097/MPA.0b013e31821bd62f. PMID 21775920
- [Background] Sahora K, Mino-Kenudson M, Brugge W, Thayer SP, Ferrone CR, Sahani D, Pitman MB, Warshaw AL, Lillemoe KD, Fernandez-del Castillo CF. Branch duct intraductal papillary mucinous neoplasms: does cyst size change the tip of the scale? A critical analysis of the revised international consensus guidelines in a large single-institutional series. Ann Surg. 2013 Sep;258(3):466-75. doi: 10.1097/SLA.0b013e3182a18f48. PMID 24022439
- [Background] Wu BU, Sampath K, Berberian CE, Kwok KK, Lim BS, Kao KT, Giap AQ, Kosco AE, Akmal YM, Difronzo AL, Yu W, Ngor EW. Prediction of malignancy in cystic neoplasms of the pancreas: a population-based cohort study. Am J Gastroenterol. 2014 Jan;109(1):121-9; quiz 130. doi: 10.1038/ajg.2013.334. Epub 2013 Oct 1. PMID 24080609
- [Background] Grobmyer SR, Cance WG, Copeland EM, Vogel SB, Hochwald SN. Is there an indication for initial conservative management of pancreatic cystic lesions? J Surg Oncol. 2009 Oct 1;100(5):372-4. doi: 10.1002/jso.21260. PMID 19267387
- [Background] Huang ES, Turner BG, Fernandez-Del-Castillo C, Brugge WR, Hur C. Pancreatic cystic lesions: clinical predictors of malignancy in patients undergoing surgery. Aliment Pharmacol Ther. 2010 Jan 15;31(2):285-94. doi: 10.1111/j.1365-2036.2009.04173.x. Epub 2009 Oct 21. PMID 19845568
- [Background] Crippa S, Bassi C, Salvia R, Malleo G, Marchegiani G, Rebours V, Levy P, Partelli S, Suleiman SL, Banks PA, Ahmed N, Chari ST, Fernandez-Del Castillo C, Falconi M. Low progression of intraductal papillary mucinous neoplasms with worrisome features and high-risk stigmata undergoing non-operative management: a mid-term follow-up analysis. Gut. 2017 Mar;66(3):495-506. doi: 10.1136/gutjnl-2015-310162. Epub 2016 Jan 7. PMID 26743012
- [Background] Springer S, Wang Y, Dal Molin M, Masica DL, Jiao Y, Kinde I, Blackford A, Raman SP, Wolfgang CL, Tomita T, Niknafs N, Douville C, Ptak J, Dobbyn L, Allen PJ, Klimstra DS, Schattner MA, Schmidt CM, Yip-Schneider M, Cummings OW, Brand RE, Zeh HJ, Singhi AD, Scarpa A, Salvia R, Malleo G, Zamboni G, Falconi M, Jang JY, Kim SW, Kwon W, Hong SM, Song KB, Kim SC, Swan N, Murphy J, Geoghegan J, Brugge W, Fernandez-Del Castillo C, Mino-Kenudson M, Schulick R, Edil BH, Adsay V, Paulino J, van Hooft J, Yachida S, Nara S, Hiraoka N, Yamao K, Hijioka S, van der Merwe S, Goggins M, Canto MI, Ahuja N, Hirose K, Makary M, Weiss MJ, Cameron J, Pittman M, Eshleman JR, Diaz LA Jr, Papadopoulos N, Kinzler KW, Karchin R, Hruban RH, Vogelstein B, Lennon AM. A combination of molecular markers and clinical features improve the classification of pancreatic cysts. Gastroenterology. 2015 Nov;149(6):1501-10. doi: 10.1053/j.gastro.2015.07.041. Epub 2015 Aug 4. PMID 26253305
- [Background] Al-Haddad MA, Kowalski T, Siddiqui A, Mertz HR, Mallat D, Haddad N, Malhotra N, Sadowski B, Lybik MJ, Patel SN, Okoh E, Rosenkranz L, Karasik M, Golioto M, Linder J, Catalano MF. Integrated molecular pathology accurately determines the malignant potential of pancreatic cysts. Endoscopy. 2015 Feb;47(2):136-42. doi: 10.1055/s-0034-1390742. Epub 2014 Oct 14. PMID 25314329
- [Background] Al-Haddad M, Wallace MB, Woodward TA, Gross SA, Hodgens CM, Toton RD, Raimondo M. The safety of fine-needle aspiration guided by endoscopic ultrasound: a prospective study. Endoscopy. 2008 Mar;40(3):204-8. doi: 10.1055/s-2007-995336. Epub 2007 Dec 4. PMID 18058615
- [Background] Boustiere C, Veitch A, Vanbiervliet G, Bulois P, Deprez P, Laquiere A, Laugier R, Lesur G, Mosler P, Nalet B, Napoleon B, Rembacken B, Ajzenberg N, Collet JP, Baron T, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Endoscopy and antiplatelet agents. European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2011 May;43(5):445-61. doi: 10.1055/s-0030-1256317. Epub 2011 May 4. PMID 21547880
- [Background] Dumonceau JM, Polkowski M, Larghi A, Vilmann P, Giovannini M, Frossard JL, Heresbach D, Pujol B, Fernandez-Esparrach G, Vazquez-Sequeiros E, Gines A; European Society of Gastrointestinal Endoscopy. Indications, results, and clinical impact of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2011 Oct;43(10):897-912. doi: 10.1055/s-0030-1256754. Epub 2011 Aug 12. PMID 21842456